CLINICAL TRIAL: NCT00986154
Title: A Phase 3, Randomized, Parallel-Group, Multi-Center, Multi-National Study for the Evaluation of Efficacy and Safety of (LMW) Heparin/Edoxaban Versus (LMW) Heparin/Warfarin in Subjects With Symptomatic Deep-Vein Thrombosis (DVT) and or Pulmonary Embolism (PE).
Brief Title: Comparative Investigation of Low Molecular Weight (LMW) Heparin/Edoxaban Tosylate (DU176b) Versus (LMW) Heparin/Warfarin in the Treatment of Symptomatic Deep-Vein Blood Clots and/or Lung Blood Clots. (The Edoxaban Hokusai-VTE Study).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DU176b-D-U305; The Edoxaban Hokusai VTE Study
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Results first posted 2015-02-25 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2015-03

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis (DVT); Pulmonary Embolism (PE); Thromboembolism; Venous Thrombosis
Keywords: Recurrent Thrombosis; Recurrent Pulmonary Embolism; Symptomatic Deep Vein Thrombosis; Symptomatic Pulmonary Embolism; Venous Thromboembolism (VTE)
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Thromboembolism; Thrombosis | interventions — edoxaban; Heparin, Low-Molecular-Weight; Heparin; Warfarin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- heparin/edoxaban tosylate (Experimental)
  Interventions: Drug: edoxaban tosylate(DU-176b); Drug: low molecular weight heparin/unfractionated heparin
- heparin/warfarin (Active Comparator)
  Interventions: Drug: low molecular weight heparin/unfractionated heparin; Drug: warfarin

INTERVENTIONS:
Drug: edoxaban tosylate(DU-176b) — edoxaban tosylate(DU-176b), film-coated tablet for oral use, 30 mg, two tablets (60 mg) once daily, maximum of 12 months treatment
  Arms: heparin/edoxaban tosylate
Drug: low molecular weight heparin/unfractionated heparin — LMW heparin - subcutaneous injection, 1 mg/Kg twice daily or 1.5 mg/Kg once daily.
  Unfractionated heparin - 5,000 IU bolus intravenous administration, 1,300 IU/hour continuous infusion, minimum of 5 days and maximum of about 12 days treatment
Drug: warfarin — tablet for oral use; 0.5 mg, 1 mg, 2.5 mg, 5 mg; daily dosage, adjusted to maintain international normalized ratio (INR) between 2.0 and 3.0; maximum of 12 months treatment
  Arms: heparin/warfarin

SUMMARY:
Evaluation of heparin/edoxaban tosylate (DU176b) versus heparin/warfarin in preventing recurrence of blood clots in patients with acute symptomatic deep-vein blood clots in the legs and/or blood clots in the lungs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects older than the minimum legal adult age (country specific);
* Acute symptomatic proximal DVT and/or symptomatic PE confirmed at the site by appropriate diagnostic imaging;
* Able to provide written informed consent

Exclusion Criteria:

* thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of DVT and/or PE;
* More than 48 hours pre-treatment with anticoagulant therapy prior to randomization;
* Calculated Creatinine clearance (CrCL) < 30 mL/min;
* significant liver disease (e.g., acute hepatitis, chronic active hepatitis, cirrhosis) or alanine transaminase (ALT) >\= 2 times the upper limit of normal (ULN), or total bilirubin (TBL) x 1.5 times the ULN;
* patients with active cancer for whom long term treatment with (LMW) heparin is anticipated;
* active bleeding or high risk for bleeding contraindicating treatment with (LMW) heparin or warfarin;
* chronic treatment with non-aspirin non-steroidal anti-inflammatory drugs (NSAIDs);
* treatment with aspirin in a dosage of more than 100 mg/per day or dual antiplatelet therapy;
* concurrent treatment with potent P-gp inhibitors;
* subjects with any condition that, as judged by the investigator, would place the subject at increased risk of harm if he/she participated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8292 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (454):
- United States (82):
  - Investigational Site 7103, Mobile, Alabama
  - Investigational Site 7132, Montgomery, Alabama
  - Investigational Site 7126, Phoenix, Arizona
  - Investigational Site 7139, Little Rock, Arkansas
  - Investigational Site 1070, Anaheim, California
  - Investigational Site 7125, Los Alamitos, California
  - Investigational Site 1093, Monterey, California
  - Investigational Site 1069, Palm Springs, California
  - Investigational Site 7150, San Diego, California
  - Investigational Site 1089, Vista, California
  - Investigational Site 1012, Aurora, Colorado
  - Investigational Site 1013, Boulder, Colorado
  - Investigational Site 1017, Denver, Colorado
  - Investigational Site 1018, Lakewood, Colorado
  - Investigational Site 1019, Littleton, Colorado
  - Investigational Site 1022, Thornton, Colorado
  - Investigational Site 1023, Thornton, Colorado
  - Brandon, Florida
  - Investigational Site 1071, Clearwater, Florida
  - Investigational Site 7117, Fort Myers, Florida
  - Investigational Site 7106, Gainesville, Florida
  - Investigational Site 1005, Ocoee, Florida
  - Investigational Site 1006, Orlando, Florida
  - Investigational Site 7144, Sarasota, Florida
  - Investigational Site 7127, St. Petersburg, Florida
  - Investigational Site 1007, Winter Park, Florida
  - Investigational Site 7104, Albany, Georgia
  - Investigational Site 1095, Columbus, Georgia
  - Investigational Site 1080, Jonesboro, Georgia
  - Investigational Site 7146, Savannah, Georgia
  - Investigational Site 1098, Park Ridge, Illinois
  - Carmel, Indiana
  - Investigational Site 7115, Paducah, Kentucky
  - Investigational Site 1065, Covington, Louisiana
  - Investigational Site 1068, Baltimore, Maryland
  - Investigational Site 1037, Westminster, Maryland
  - Investigational Site 1038, Westminster, Maryland
  - Investigational Site 7133, Kansas City, Missouri
  - Investigational Site 7147, Butte, Montana
  - Investigational Site 1039, Las Vegas, Nevada
  - Investigational Site 7143, Rochester, New York
  - Investigational Site 7135, Durham, North Carolina
  - Investigational Site 7145, Statesville, North Carolina
  - Investigational Site 7138, Maumee, Ohio
  - Investigational Site 7122, Toledo, Ohio
  - Investigational Site 7152, Bend, Oregon
  - Portland, Oregon
  - Investigational Site 1004, Camp Hill, Pennsylvania
  - Investigational Site 7109, Ephrata, Pennsylvania
  - Investigational Site 1049, Kingston, Pennsylvania
  - Investigational Site 7109, Lancaster, Pennsylvania
  - Investigational Site 7154, Sellersville, Pennsylvania
  - Investigational Site 7128, Uniontown, Pennsylvania
  - Investigational Site 1031, Easley, South Carolina
  - Investigational Site 1032, Greenville, South Carolina
  - Investigational Site 1034, Greenville, South Carolina
  - Investigational Site 1033, Greenville, South Carolina
  - Investigational Site 1035, Seneca, South Carolina
  - Investigational Site 1036, Spartanburg, South Carolina
  - Investigational Site 1009, Arlington, Texas
  - Investigational Site 1050, Dallas, Texas
  - Investigational Site 1047, Fort Worth, Texas
  - Investigational Site 7105, Fort Worth, Texas
  - Investigational Site 1048, Fort Worth, Texas
  - Investigational Site 1059, Midland, Texas
  - Investigational Site 1040, New Braunfels, Texas
  - Investigational Site 1041, Odessa, Texas
  - Investigational Site 1002, San Antonio, Texas
  - Investigational Site 1058, Sugar Land, Texas
  - Investigational Site 1042, Tyler, Texas
  - Investigational Site 1008, Waco, Texas
  - Investigational Site 7123, Salt Lake City, Utah
  - Investigational Site 1003, Fredericksburg, Virginia
  - Investigational Site 1025, Newport News, Virginia
  - Investigational Site 1024, Norfolk, Virginia
  - Investigational Site 1066, Randallstown, Virginia
  - Investigational Site 1030, Virginia Beach, Virginia
  - Investigational Site 7120, Seattle, Washington
  - Investigational Site 1076, Tacoma, Washington
  - Investigational Site 1053, Vancouver, Washington
  - Investigational Site 1056, Vancouver, Washington
  - Investigational Site 1057, Vancouver, Washington
- Argentina (7):
  - Investigational Site 1100, Buenos Aires
  - Investigational Site 1103, Buenos Aires
  - Investigational Site 1106, Buenos Aires
  - Investigational Site 1108, Buenos Aires
  - Investigational Site 1104, Córdoba
  - Investigational Site 1110, Pcia de Corrientes
  - Investigational Site 1109, Santa Fe
- Australia (12):
  - Investigational Site 4205, Bedford Park
  - Investigational Site 4209, Box Hill
  - Investigational Site 4210, Clayton
  - Investigational Site 4211, Fremantle
  - Investigational Site 4213, Garran
  - Kogarah
  - Investigational Site 4207, Perth
  - Investigational Site 4203, Redcliffe
  - Investigational Site 4206, Saint Leonards NSW
  - Investigational Site 4214, South Brisbane
  - Investigational Site 4212, Westmead NSW
  - Investigational Site 4200, Windsor
- Austria (6):
  - Investigational Site 2802, Feldkirch
  - Investigational Site 2803, Graz
  - Investigational Site 2800, Innsbruck
  - Investigational Site 2804, Linz
  - Sr. M. Restitutagasse
  - Vienna
- Belarus (6):
  - Investigational Site 2704, Grodno
  - Investigational Site 2703, Homyel
  - Investigational Site 2700, Minsk
  - Investigational site 2701, Minsk
  - Investigational Site 2702, Minsk
  - Investigational Site 2705, Mogilev
- Belgium (2):
  - Investigational Site 1608, Aalst
  - Investigational Site 1602, Lier
- Brazil (13):
  - Investigational Site 2905, Belo Horizonte
  - Investigational Site 2914, Campinas
  - Investigational Site 2901, Curitiba
  - Investigational Site 2903, Curitiba
  - Investigational Site 2912, Porto Alegre
  - Investigational Site 2915, Porto Alegre
  - Investigational Site 2917, Porto Alegre
  - Investigational Site 2904, São Bernardo do Campo
  - Investigational Site 2900, São Paulo
  - Investigational Site 2902, São Paulo
  - Investigational Site 2906, São Paulo
  - Investigational Site 2910, São Paulo
  - Investigational Site 2911, São Paulo
- Canada (7):
  - Investigational Site 2006, Edmonton, Alberta
  - Investigational Site 2001, London, Ontario
  - Investigational Site 2007, Newmarket, Ontario
  - Investigational Site 2000, Ottawa, Ontario
  - Investigational Site 2003, Richmond Hill, Ontario
  - Investigational Site 2005, Halifax
  - Investigational Site 2004, Montreal
- Chile (2):
  - Investigational Site 1200, Santiago
  - Investigational Site 1204, Santiago
- China (24):
  - Investigational Site 4301, Beijing
  - Investigational Site 4302, Beijing
  - Investigational Site 4306, Beijing
  - Investigational Site 4321, Beijing
  - Investigational Site 4327, Beijing
  - Investigational Site 4337, Beijing
  - Investigational Site 4316, Guangzhou
  - Investigational Site 4310, Hangzhou
  - Hebei Province
  - Investigational Site 4325, Jiangsu
  - Investigational Site 4317, Kunming
  - Investigational Site 4328, Nanjing
  - Investigational Site 4319, Nanning
  - Investigational Site 4313, Qingdao
  - Investigational Site 4303, Shanghai
  - Investigational Site 4324, Shanghai
  - Investigational Site 4330, Shanghai
  - Investigational Site 4335, Shanghai
  - Investigational Site 4326, Shenyang
  - Investigational Site 4308, Sichuan Province
  - Investigational Site 4318, Taiyuan
  - Investigational Site 4320, Tianjin
  - Investigational site 4338, Xi'an
  - Investigational Site 4315, Yinchuan
- Czechia (9):
  - Chodov
  - Jihlava
  - Investigational Site 1902, Liberec
  - Investigational Site 1908, Olomouc
  - Investigational Site 1905, Ostrava
  - Investigational Site 1901, Pilsen
  - Investigational Site 1910, Pilsen
  - Investigational Site 1904, Prague
  - Ústí nad Labem
- Denmark (6):
  - Investigational Site 6010, Aarhus
  - Arhus N.
  - Copenhagen
  - Investigational Site 6003, Herlev
  - Ringvej
  - Investigational Site 6001, Svendborg
- Estonia (3):
  - Investigational Site 2100, Tallinn
  - Investigational Site 2101, Tallinn
  - Investigational Site 2102, Tartu
- France (32):
  - Investigational Site 3314, Agen
  - Investigational Site 3302, Amiens
  - Investigational Site 3311, Angers
  - Investigational Site 3321, Annecy
  - Investigational Site 3300, Arras
  - Investigational Site 3301, Besançon
  - Investigational Site 3329, Bordeaux
  - Investigational Site 3310, Brest
  - Investigational Site 3333, Cannes
  - Investigational Site 3327, Colombes
  - Investigational Site 3323, Dijon
  - Investigational Site 3307, Grenoble
  - Investigational Site 3322, Grenoble
  - Investigational Site 3325, Hetztessy
  - Investigational Site 3328, Le Mans
  - Investigational Site 3339, Lille
  - Lormont
  - Investigational Site 3318, Lyon
  - Investigational Site 3303, Montpellier
  - Nantes
  - Investigational Site 3319, Nice
  - Investigational Site 3308, Paris
  - Investigational Site 3312, Paris
  - Investigational Site 3313, Paris
  - Investigational Site 3337, Paris
  - Investigational Site 3335, Pessac
  - Investigational Site 3341, Pessac
  - Investigational Site 3336, Pierre-Bénite
  - Roskilde
  - Saint Aubin Surscie
  - Investigational Site 3305, Saint-Etienne
  - Investigational Site 3316, Toulon
- Germany (15):
  - Investigational Site 1718, Berlin
  - Investigational Site 1720, Bielefeld
  - Investigational Site 1715, Bruchsal
  - Investigational Site 1700, Darmstadt
  - Investigational Site 1719, Dortmund
  - Investigational Site 1701, Dresden
  - Investigational Site 1707, Dresden
  - Investigational Site 1721, Hamburg
  - Magdeburg
  - Investigational Site 1712, Mainz
  - Investigational Site 1704, München
  - Investigational Site 1714, Nordhausen
  - Investigational Site 1711, Paderborn
  - Investigational Site 1706, Tübingen
  - Investigational Site 1708, Witten
- Hungary (16):
  - Investigational Site 5413, Baja
  - Investigational Site 5401, Budapest
  - Investigational Site 5404, Budapest
  - Investigational Site 5409, Budapest
  - Investigational Site 5414, Budapest
  - Investigational Site 5400, Debrecen
  - Investigational Site 5402, Kecskemét
  - Investigational Site 5405, Kistarcsa
  - Maglodi
  - Investigational Site 5407, Miskolc
  - Investigational Site 5410, Pécs
  - Rakoczi
  - Investigational Site 5403, Szentes
  - Investigational Site 5408, Szombathely
  - Investigational Site 5412, Zalaegerszeg
  - Zrinyi
- India (37):
  - Ahmedabad
  - Andhra Pradesh
  - Investigational Site 4402, Bangalore
  - Investigational Site 4405, Bangalore
  - Investigational Site 4442, Bangalore
  - Investigational Site 4459, Bangalore
  - Investigational Site 4460, Bangalore
  - Investigational Site 4472, Bangalore
  - Gujarat
  - Gūrgaon
  - Haryāna
  - Investigational Site 5514, Holon
  - Investigational Site 4407, Hyderabad
  - Investigational Site 4430, Hyderabad
  - Investigational Site 4444, Hyderabad
  - Investigational Site 4451, Hyderabad
  - Karnataka
  - Kerala
  - Investigational Site 4420, Lucknow
  - Madhya Pradesh
  - Maharashtra
  - Investigational Site 4409, Mumbai
  - Investigational Site 4424, Mumbai
  - Investigational Site 4419, New Delhi
  - Investigational Site 4428, New Delhi
  - Investigational Site 4441, New Delhi
  - Investigational Site 4425, Pune
  - Investigational Site 4438, Pune
  - Investigational Site 4443, Pune
  - Investigational Site 4462, Pune
  - Punjab
  - Rajasthan
  - Investigational Site 4470, Secunderbad
  - Tamil Nadu
  - Uttar Pradesh
  - Vadodara
  - Visakhapatnam
- Israel (13):
  - Afula
  - Ashkelon
  - Hadera
  - Investigational Site 5506, Haifa
  - Investigational Site 5508, Haifa
  - Investigational Site 5500, Holon
  - Investigational Site 5501, Jerusalem
  - Investigational Site 5505, Kfar Saba
  - Investigational Site 5513, Nahariya
  - Investigational Site 5510, Petah Tikva
  - Investigational Site 5512, Poria – Neve Oved
  - Investigational Site 5503, Tel Aviv
  - Investigational Site 5509, Tel Litwinsky
- Italy (12):
  - Investigational Site 3508, Bergamo
  - Investigational Site 3506, Chieti
  - Investigational Site 3500, Emilia
  - Investigational Site 3504, Milan
  - Padua
  - Investigational Site 3502, Palermo
  - Investigational Site 3507, Parma
  - Investigational Site 3501, Pavia
  - Investigational Site 3505, Rozzano
  - Investigational Site 3510, Udine
  - Investigational Site 3503, Varese
  - Investigational Site 3509, Venezia
- Japan (32):
  - Investigational Site 6137, Aichi
  - Investigational Site 6104, Aomori
  - Investigational Site 6117, Chiba
  - Investigational Site 6119, Fukuoka
  - Fukuoka
  - Investigational Site 6110, Fukushima
  - Investigational Site 6150, Hiroshima
  - Investigational Site 6138, Hokkaido
  - Investigational Site 6141, Hokkaido
  - Investigational Site 6133, Hyōgo
  - Hyōgo
  - Investigational Site 6114, Ishikawa
  - Investigational Site 6144, Kagoshima
  - Investigational Site 6112, Kanagawa
  - Investigational Site 6123, Kumamoto
  - Investigational Site 6147, Kumamoto
  - Investigational Site 6148, Kumamoto
  - Investigational Site 6129, Mie
  - Investigational Site 6146, Nagano
  - Investigational Site 6139, Nagasaki
  - Investigational Site 6107, Niigata
  - Investigational Site 6152, Okayama
  - Investigational Site 6135, Okinawa
  - Investigational Site 6132, Osaka
  - Investigational Site 6130, Sapporo
  - Investigational Site 6143, Shizuoka
  - Investigational Site 6102, Tokyo
  - Investigational Site 6105, Tokyo
  - Investigational Site 6113, Tokyo
  - Investigational Site 6142, Tokyo
  - Investigational Site 6145, Tokyo
  - Investigational Site 6149, Tottori
- Mexico (9):
  - Investigational Site 1303, Zapopan, Jalisco
  - Investigational Site 1302, Monterrey, Nuevo León
  - Investigational Site 1311, Col. Lomas Altas C.P
  - Investigational Site 1304, Guadalajara
  - Investigational Site 1312, Guadalajara
  - Investigational Site 1300, Hermosillo
  - Investigational Site 1305, Monterrey, Nuevo Leon
  - Investigational Site 1308, San Luis Potosí City
  - Investigational Site 1301, Yucatán
- Netherlands (10):
  - Investigational Site 3608, Alkmaar
  - Investigational Site 3607, Almere Stad
  - Investigational Site 3617, Amersfoort
  - Investigational Site 3611, Amsterdam
  - Investigational Site 3609, Assen
  - Investigational Site 3603, Groningen
  - Investigational Site 3612, Heerlen
  - Investigational Site 3613, Hoofddorp
  - Investigational Site 3602, Nijmegen
  - Investigational Site 3615, Rotterdam
- New Zealand (4):
  - Investigational Site 4702, Auckland
  - Investigational Site 4703, Auckland
  - Investigational Site 4700, Christchurch
  - Investigational Site 4704, Wellington
- Norway (2):
  - Investigational Site 3701, Fredrikstad
  - Investigational Site 3700, Oslo
- Philippines (4):
  - Pasig
  - Investigational Site 4800, Quezon City
  - Investigational site 4801, Quezon City
  - Investigational Site 4802, Quezon City
- Poland (8):
  - Investigational Site 5015, Bialystok
  - Investigational Site 5005, Krakow
  - Investigational Site 5019, Olsztyn
  - Investigational Site 5018, Tarnów
  - Investigational Site 5003, Warsaw
  - Investigational Site 5007, Warsaw
  - Investigational Site 5008, Warsaw
  - Investigational Site 5014, Warsaw
- Russia (19):
  - Barnaul
  - Investigational Site 3023, Chelyabinsk
  - Investigational Site 3017, Irkutsk
  - Investigational Site 3019, Kemerovo
  - Investigational Site 3020, Krasnoyarsk
  - Investigational Site 3030, Krasnoyarsk
  - Investigational Site 3029, Moscow
  - Investigational Site 3028, Novosibirsk
  - Investigational Site 3009, Omsk
  - Investigational Site 3022, Ryazan
  - Investigational Site 3000, Saint Petersburg
  - Investigational Site 3003, Saint Petersburg
  - Investigational Site 3027, Saint Petersburg
  - Saratov
  - Investigational Site 3024, Sochi
  - Investigational Site 3025, Tyumen
  - Investigational Site 3016, Ufa
  - Investigational Site 3004, Yaroslavl
  - Investigational Site 3010, Yaroslavl
- Singapore (2):
  - Investigational Site 5900, Outram Road
  - Investigational Site 5902, Singapore
- South Africa (11):
  - Investigational Site 4912, Cape Town
  - Investigational Site 4907, Centurion
  - Investigational Site 4901, Johannesburg
  - Investigational Site 4905, Johannesburg
  - Investigational Site 4909, Johannesburg
  - Investigational Site 4910, Johannesburg
  - Investigational Site 4908, Lyttleton
  - Investigational Site 4903, Pretoria
  - Investigational Site 4906, Pretoria
  - Investigational Site 4904, Somerset West
  - Investigational Site 4900, Worcester
- South Korea (7):
  - Investigational Site 4513, Busan
  - Investigational Site 4509, Daegu
  - Investigational Site 4501, Gyeonggi-do
  - Investigational Site 4506, Seoul
  - Investigational Site 4507, Seoul
  - Investigational Site 4508, Seoul
  - Investigational Site 4515, Seoul
- Spain (2):
  - Investigational site 1503, Barcelona
  - Investigational Site 1502, Cabra
- Sweden (5):
  - Investigational Site 3900, Hällingsjö
  - Investigational Site 3904, Kristianstad
  - Investigational Site 3903, Stockholm
  - Investigational Site 3905, Stockholm
  - Investigational Site 3902, Sundsvall
- Switzerland (6):
  - Investigational Site 4103, Aarau
  - Investigational Site 4110, Basel
  - Investigational Site 4104, Bellinzona
  - Investigational Site 4102, Chur
  - Investigational Site 4109, Lausanne
  - Investigational Site 4100, Lucerne
- Taiwan (5):
  - Hualien City
  - Investigational Site 5104, Kaohsiung City
  - Investigational Site 5105, Taichung
  - Investigational Site 5101, Taipei
  - Investigational Site 5103, Taipei
- Thailand (3):
  - Investigational Site 5200, Bangkok
  - Investigational Site 5202, Bangkok
  - Investigational Site 5203, Nakhorn Nayok
- Turkey (Türkiye) (4):
  - Investigational Site 5702, Ankara
  - Investigational Site 5703, Ankara
  - Investigational Site 5702, Istanbul
  - Investigational Site 5706, Istanbul
- Ukraine (10):
  - Chernihiv
  - Investigational Site 4008, Dnipropetrovsk
  - Investigational Site 4010, Donetsk
  - Investigational Site 4000, Ivano-Frankivsk
  - Investigational Site 4002, Kharkiv
  - Investigational Site 4001, Kiev
  - Investigational Site 4007, Ternopil
  - Investigational Site 4009, Uzhhorod
  - Investigational Site 4003, Vinnitsya
  - Investigational Site 4006, Zaporizhzhia
- United Kingdom (7):
  - Investigational Site 7005, Coventry
  - Investigational Site 7006, Hull
  - Investigational Site 7000, London
  - Investigational Site 7003, London
  - Investigational Site 7004, London
  - Investigational Site 7001, Newcastle
  - Investigational Site 7007, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Christodoulou KC, Barco S, Abele C, Lodigiani C, Monreal M, Konstantinides SV, Valerio L. Burden of Atherosclerosis and Outcomes of Acute Pulmonary Embolism: A Post Hoc Analysis of the Hokusai-VTE Trial. J Am Heart Assoc. 2025 Nov 18;14(22):e041420. doi: 10.1161/JAHA.125.041420. Epub 2025 Nov 6. PMID 41195787
- [Derived] Vanassche T, Verhamme P, Wells PS, Segers A, Ageno W, Brekelmans MPA, Chen CZ, Cohen AT, Grosso MA, Medina AP, Mercuri MF, Winters SM, Zhang G, Weitz JI, Raskob GE, Buller HR. Impact of age, comorbidity, and polypharmacy on the efficacy and safety of edoxaban for the treatment of venous thromboembolism: An analysis of the randomized, double-blind Hokusai-VTE trial. Thromb Res. 2018 Feb;162:7-14. doi: 10.1016/j.thromres.2017.12.005. Epub 2017 Dec 13. PMID 29248859
- [Derived] Vandell AG, Walker J, Brown KS, Zhang G, Lin M, Grosso MA, Mercuri MF. Genetics and clinical response to warfarin and edoxaban in patients with venous thromboembolism. Heart. 2017 Nov;103(22):1800-1805. doi: 10.1136/heartjnl-2016-310901. Epub 2017 Jul 8. PMID 28689179
- [Derived] Brekelmans MP, Ageno W, Beenen LF, Brenner B, Buller HR, Chen CZ, Cohen AT, Grosso MA, Meyer G, Raskob G, Segers A, Vanassche T, Verhamme P, Wells PS, Zhang G, Weitz JI. Recurrent venous thromboembolism in patients with pulmonary embolism and right ventricular dysfunction: a post-hoc analysis of the Hokusai-VTE study. Lancet Haematol. 2016 Sep;3(9):e437-45. doi: 10.1016/S2352-3026(16)30080-1. PMID 27570090
- [Derived] Raskob GE, van Es N, Segers A, Angchaisuksiri P, Oh D, Boda Z, Lyons RM, Meijer K, Gudz I, Weitz JI, Zhang G, Lanz H, Mercuri MF, Buller HR; Hokusai-VTE investigators. Edoxaban for venous thromboembolism in patients with cancer: results from a non-inferiority subgroup analysis of the Hokusai-VTE randomised, double-blind, double-dummy trial. Lancet Haematol. 2016 Aug;3(8):e379-87. doi: 10.1016/S2352-3026(16)30057-6. Epub 2016 Jul 1. PMID 27476789
- [Derived] Nakamura M, Wang YQ, Wang C, Oh D, Yin WH, Kimura T, Miyazaki K, Abe K, Mercuri M, Lee LH, Segers A, Buller H. Efficacy and safety of edoxaban for treatment of venous thromboembolism: a subanalysis of East Asian patients in the Hokusai-VTE trial. J Thromb Haemost. 2015 Sep;13(9):1606-14. doi: 10.1111/jth.13055. Epub 2015 Aug 27. PMID 26179767
- [Derived] Hokusai-VTE Investigators; Buller HR, Decousus H, Grosso MA, Mercuri M, Middeldorp S, Prins MH, Raskob GE, Schellong SM, Schwocho L, Segers A, Shi M, Verhamme P, Wells P. Edoxaban versus warfarin for the treatment of symptomatic venous thromboembolism. N Engl J Med. 2013 Oct 10;369(15):1406-15. doi: 10.1056/NEJMoa1306638. Epub 2013 Aug 31. PMID 23991658
- [Derived] Camm AJ, Bounameaux H. Edoxaban: a new oral direct factor xa inhibitor. Drugs. 2011 Aug 20;71(12):1503-26. doi: 10.2165/11595540-000000000-00000. PMID 21861537

RESULTS

PARTICIPANT FLOW:
Groups:
- Heparin/Edoxaban Tosylate: edoxaban tosylate(DU-176b): edoxaban tosylate(DU-176b), film-coated tablet for oral use, 30 mg, two tablets (60 mg) once daily, maximum of 12 months treatment
  low molecular weight heparin/unfractionated heparin: LMW heparin - subcutaneous injection, 1 mg/Kg twice daily or 1.5 mg/Kg once daily.
  Unfractionated heparin - 5,000 IU bolus intravenous administration, 1,300 IU/hour continuous infusion, minimum of 5 days and maximum of about 12 days treatment
- Heparin/Warfarin: low molecular weight heparin/unfractionated heparin: LMW heparin - subcutaneous injection, 1 mg/Kg twice daily or 1.5 mg/Kg once daily.
  Unfractionated heparin - 5,000 IU bolus intravenous administration, 1,300 IU/hour continuous infusion, minimum of 5 days and maximum of about 12 days treatment
  warfarin: tablet for oral use; 0.5 mg, 1 mg, 2.5 mg, 5 mg; daily dosage, adjusted to maintain international normalized ratio (INR) between 2.0 and 3.0; maximum of 12 months treatment
Period: Overall Study
Arm/Group | Heparin/Edoxaban Tosylate | Heparin/Warfarin
Started | 4143 | 4149
Safety Analysis Set (Received Drug) | 4118 | 4122
Completed | 3937 | 3955
Not Completed | 206 | 194
Not completed — Death | 136 | 127
Not completed — Lost to Follow-up | 7 | 4
Not completed — Withdrawal by Subject | 32 | 33
Not completed — investigator/subject decide not continue | 6 | 3
Not completed — never received study drug | 25 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heparin/Edoxaban Tosylate | Heparin/Warfarin | Total
Number analyzed (Participants) | 4118 | 4122 | 8240
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (16.3) | 55.9 (16.2) | 55.8 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1758 | 1766 | 3524
  Male | 2360 | 2356 | 4716
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 866 | 861 | 1727
  Native Hawaiian or Other Pacific Islander | 0 | 4 | 4
  Black or African American | 156 | 144 | 300
  White | 2867 | 2895 | 5762
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 229 | 218 | 447
Region of Enrollment [Number; unit: participants]
  Belarus | 40 | 44 | 84
  United States | 307 | 311 | 618
  Philippines | 17 | 15 | 32
  Taiwan | 74 | 64 | 138
  Estonia | 40 | 36 | 76
  Thailand | 18 | 24 | 42
  Spain | 19 | 8 | 27
  Ukraine | 143 | 148 | 291
  Russian Federation | 260 | 257 | 517
  Israel | 106 | 125 | 231
  Switzerland | 27 | 20 | 47
  Italy | 70 | 83 | 153
  India | 245 | 266 | 511
  France | 364 | 350 | 714
  Denmark | 123 | 143 | 266
  Australia | 90 | 89 | 179
  South Africa | 185 | 180 | 365
  Netherlands | 188 | 197 | 385
  China | 243 | 241 | 484
  Korea, Republic of | 140 | 130 | 270
  Turkey | 27 | 24 | 51
  Austria | 80 | 86 | 166
  United Kingdom | 44 | 67 | 111
  Czech Republic | 216 | 211 | 427
  Hungary | 230 | 232 | 462
  Mexico | 59 | 67 | 126
  Canada | 109 | 109 | 218
  Argentina | 26 | 21 | 47
  Poland | 22 | 21 | 43
  Brazil | 46 | 44 | 90
  Belgium | 98 | 79 | 177
  Singapore | 7 | 4 | 11
  Norway | 15 | 15 | 30
  Germany | 243 | 230 | 473
  Japan | 106 | 103 | 209
  New Zealand | 55 | 56 | 111
  Sweden | 36 | 22 | 58

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Recurrent VTE, i.e., the Composite of DVT, Non-fatal PE, and Fatal PE
Description: Symptomatic recurrent Venous Thromboembolism (VTE), i.e., the composite of deep Vein Thrombosis (DVT), non-fatal Pulmonary Embolism (PE), and fatal PE occurring during the Overall Study Period.
  Overall Study Period defined as "The time from the reference date (randomization date/initial dose of study drug date) to the last study follow-up visit."
Time Frame: 12 months from time of randomization
Population: (mITT) modified Intent To Treat Analysis Set
Measure: Number; unit: number or participants with an event
Arm/Group | Heparin/Edoxaban Tosylate | Heparin/Warfarin
Number analyzed (Participants) | 4118 | 4122
number or participants with an event | 130 | 146
Statistical Analysis 1: Comparison: Heparin/Edoxaban Tosylate vs Heparin/Warfarin; (LMW) heparin/edoxaban will be non-inferior to (LMW) heparin/warfarin in preventing recurrence of acute, symptomatic VTE following initial index event. (LMW) Heparin/edoxaban was considered non-inferior to the standard therapy ([LMW] heparin/warfarin) if the upper limit of the two-sided 95% confidence interval (CI) for the Hazard Ratio ([LMW] heparin/edoxaban to standard therapy) was less than 1.5. Events included in Overall study period if occurred on or after randomization date up to Day 365; Test type: Non-Inferiority or Equivalence — The study was designed to accumulate approximately 220 Overall primary efficacy events in the mITT (modified Intent to Treat) Analysis Set. Assuming equal efficacy (Hazard Ratio = 1.00), a total of 220 events gave a power of 85% to demonstrate that (LMW) heparin/edoxaban was non-inferior to the comparator, considering a relative non-inferiority margin of 1.5 (two sided α=0.05); p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [.703 to 1.128] — Time to 1st event analyzed by Cox proportional hazards with terms treatment group, randomization stratification factors: Presenting Diagnosis (PE with/without DVT, DVT only); Baseline risk factors (temp factors; all others); Need for reduced dose

2. Secondary Outcome: The Composite Clinical Outcome of Symptomatic Recurrent VTE and All-cause Mortality
Time Frame: 12 months from time of randomization
Population: mITT Analysis set
Measure: Number; unit: number of participants with event
Arm/Group | Heparin/Edoxaban Tosylate | Heparin/Warfarin
Number analyzed (Participants) | 4118 | 4122
number of participants with event | 228 | 228
Statistical Analysis 1: Comparison: Heparin/Edoxaban Tosylate vs Heparin/Warfarin; Test type: Superiority or Other; p = .9933, Regression, Cox; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [.832 to 1.200] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Clinically Relevant Bleeding (i.e., Major or Clinically Relevant Non-major Bleeding) Occurring During Treatment
Description: Clinically relevant bleeding (i.e., major or clinically relevant non-major bleeding) occurring during treatment plus 3 days after their last dose for that time period.
Time Frame: 12 months from time of randomization
Population: Safety Analysis Set
Measure: Number; unit: participants with an event
Arm/Group | Heparin/Edoxaban Tosylate | Heparin/Warfarin
Number analyzed (Participants) | 4118 | 4122
participants with an event | 349 | 423
Statistical Analysis 1: Comparison: Heparin/Edoxaban Tosylate vs Heparin/Warfarin; Safety Analysis set includes all randomized subjects who received at least one dose of study drug. Null hypothesis (LMW) heparin/edoxaban will be comparable to (LMW) heparin/warfarin in preventing recurrence of major or clinically relevant non-major bleeding; Test type: Superiority or Other; p = .0040, Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [.705 to .936] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Heparin/Edoxaban Tosylate | Heparin/Warfarin
Serious Adverse Events (participants affected / at risk) | 801/4118 | 852/4122
Other Adverse Events (participants affected / at risk) | 816/4118 | 997/4122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heparin/Edoxaban Tosylate (N=4118) | Heparin/Warfarin (N=4122)
Pneumonia (Infections and infestations) | 35 (36) | 31 (32)
Sepsis (Infections and infestations) | 13 (13) | 10 (10)
Urinary tract infection (Infections and infestations) | 11 (12) | 11 (11)
Bronchitis (Infections and infestations) | 10 (10) | 3 (3)
Septic shock (Infections and infestations) | 8 (8) | 5 (5)
Cellulitis (Infections and infestations) | 7 (8) | 13 (15)
Diverticulitis (Infections and infestations) | 4 (4) | 1 (1)
Bronchopneumonia (Infections and infestations) | 3 (3) | 2 (2)
Erysipelas (Infections and infestations) | 3 (4) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Abdominal abscess (Infections and infestations) | 2 (2) | 1 (2)
Lobar pneumonia (Infections and infestations) | 2 (2) | 2 (3)
Lung infection (Infections and infestations) | 2 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 0 (0)
AIDS related complication (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 4 (4)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Coxsackie viral infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (2) | 0 (0)
Periorbital abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (2)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 2 (3)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 2 (2)
Cystitis escherichia (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus hepatitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 2 (2)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (3)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Gingival abscess (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1)
Implant site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Infected bites (Infections and infestations) | 0 (0) | 1 (1)
Infectious peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pancreatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (5)
Septic phlebitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Splenic abscess (Infections and infestations) | 0 (0) | 1 (2)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Testicular abscess (Infections and infestations) | 0 (0) | 1 (1)
Thrombophlebitis septic (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral myocarditis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 3 (3)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 8 (8)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 7 (7)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 8 (8)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (4)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 3 (3)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (5) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Genitourinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Inflammatory myofibroblastic tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 13 (14)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenocyst (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pernicious anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypocoagulable state (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Behcet's syndrome (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Polyarteritis nodosa (Immune system disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 4 (4)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (5)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 3 (3)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 12 (12) | 7 (8)
Syncope (Nervous system disorders) | 11 (12) | 5 (5)
Cerebral infarction (Nervous system disorders) | 6 (6) | 3 (3)
Ischaemic stroke (Nervous system disorders) | 5 (6) | 5 (6)
Headache (Nervous system disorders) | 4 (4) | 4 (5)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 8 (8)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 2 (2)
Paraplegia (Nervous system disorders) | 2 (2) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 7 (7)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Complicated migraine (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Drug withdrawal headache (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (3) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lower motor neurone lesion (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (2) | 6 (7)
Senile dementia (Nervous system disorders) | 1 (1) | 0 (0)
Spinal vascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Brown-Sequard syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 2 (2)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 5 (8)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (2) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 5 (5)
Myocardial infarction (Cardiac disorders) | 17 (18) | 7 (7)
Cardiac failure (Cardiac disorders) | 14 (18) | 7 (8)
Atrial fibrillation (Cardiac disorders) | 11 (11) | 3 (3)
Angina pectoris (Cardiac disorders) | 5 (5) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 12 (12)
Cardiac arrest (Cardiac disorders) | 4 (4) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 10 (13)
Angina unstable (Cardiac disorders) | 3 (4) | 4 (4)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 2 (2) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (2)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 2 (4)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale chronic (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 4 (4)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Eosinophilic myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 4 (4)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 2 (2)
Dressler's syndrome (Cardiac disorders) | 0 (0) | 1 (2)
Hypertensive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 2 (2)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 43 (43) | 70 (72)
Arteriosclerosis (Vascular disorders) | 4 (4) | 0 (0)
Haematoma (Vascular disorders) | 4 (5) | 16 (17)
Hypertensive crisis (Vascular disorders) | 4 (4) | 2 (2)
Aortic aneurysm (Vascular disorders) | 3 (3) | 0 (0)
Venous insufficiency (Vascular disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Post thrombotic syndrome (Vascular disorders) | 2 (2) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 2 (2)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 1 (1)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhagic infarction (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
May-Thurner syndrome (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0)
Vascular occlusion (Vascular disorders) | 1 (2) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 0 (0) | 1 (2)
Intra-abdominal haematoma (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Necrosis ischaemic (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 64 (64) | 69 (73)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 6 (6)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 (18) | 14 (16)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (8)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 15 (18) | 12 (12)
Rectal haemorrhage (Gastrointestinal disorders) | 11 (11) | 9 (9)
Pancreatitis (Gastrointestinal disorders) | 6 (9) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (6) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Melaena (Gastrointestinal disorders) | 2 (2) | 4 (4)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Volvulus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal erosion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhagic ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ileal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal strangulation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatolithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 2 (2)
Sigmoiditis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 6 (6) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 3 (3)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haemobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cytolytic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis fulminant (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Finger deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CREST syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 12 (13) | 25 (25)
Renal failure acute (Renal and urinary disorders) | 8 (8) | 7 (8)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 3 (3)
Urinary retention (Renal and urinary disorders) | 3 (3) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 2 (2)
Nephropathy toxic (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Bladder hypertrophy (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder mass (Renal and urinary disorders) | 1 (1) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 2 (2)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral meatus stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 9 (10) | 3 (3)
Vaginal haemorrhage (Reproductive system and breast disorders) | 5 (5) | 5 (6)
Menometrorrhagia (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Uterine haemorrhage (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterine mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vaginal lesion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Polymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Premenstrual syndrome (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haemangioma congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 18 (19) | 10 (11)
Death (General disorders) | 10 (10) | 9 (9)
Non-cardiac chest pain (General disorders) | 8 (8) | 6 (6)
Oedema peripheral (General disorders) | 7 (7) | 4 (4)
Multi-organ failure (General disorders) | 3 (3) | 2 (2)
Device dislocation (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Inflammation (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 2 (2) | 4 (4)
Sudden death (General disorders) | 2 (2) | 2 (2)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0)
Device leakage (General disorders) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (2) | 0 (0)
Granuloma (General disorders) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0)
Metaplasia (General disorders) | 1 (1) | 0 (0)
Multi-organ disorder (General disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 6 (7)
Accidental death (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (2)
Therapeutic response increased (General disorders) | 0 (0) | 1 (1)
Thrombosis in device (General disorders) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 12 (13) | 79 (89)
Hepatic enzyme increased (Investigations) | 5 (5) | 3 (3)
Liver function test abnormal (Investigations) | 2 (2) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Coagulation test abnormal (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 1 (1)
Pulmonary arterial pressure increased (Investigations) | 1 (1) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1)
Smear cervix abnormal (Investigations) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 7 (7) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 5 (5) | 7 (7)
Joint dislocation (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Spinal compression fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Operative haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 4 (5)
Failure to anastomose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Abortion induced (Surgical and medical procedures) | 3 (3) | 4 (4)
Prosthesis user (Social circumstances) | 1 (1) | 0 (0)
Homicide (Social circumstances) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heparin/Edoxaban Tosylate (N=4118) | Heparin/Warfarin (N=4122)
nasopharyngitis (Infections and infestations) | 260 (319) | 254 (316)
headache (Nervous system disorders) | 248 (291) | 208 (287)
pain in extremity (Musculoskeletal and connective tissue disorders) | 235 (276) | 218 (241)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 208 (263) | 246 (353)
international normalised ratio increased (Investigations) | 27 (33) | 275 (386)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A study site may not publish results of a study until after a coordinated multicenter publication has been submitted for publication or until one year after the study has ended, whichever occurs first. The study site will have the opportunity to publish results of the study, provided Daiichi Sankyo has had the opportunity to review and comment on the study site's proposed publication prior to being submitted for publication with the advice of patent council and need for subject protection.